CLINICAL TRIAL: NCT03079557
Title: A Non-randomised, Open Feasibility Pilot for the 'REpurposing BOtulinum Toxin in Treatment of Obesity in Adolescents' (ReBOO) Trial
Brief Title: Feasibility Pilot for the ReBOO-trial
Acronym: ReBOO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESA 17/1878; 2016-000326-19 (EudraCT Number)
Record Dates: First submitted 2017-02-26; First posted 2017-03-14 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Obesity
Keywords: Adolescent; Injections, intraperitoneal; Endoscopy; Botulinum Toxins, Type A; OnabotulinumtoxinA
MeSH Terms: conditions — Obesity | interventions — Idoxuridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intragastric botulinum toxin type A (Experimental): Botulinum toxin A (Allergan) injected intragastrically in the antrum
  Interventions: Drug: Intragastric botulinum toxin type A

INTERVENTIONS:
Drug: Intragastric botulinum toxin type A — 200 units Botulinum toxin A (Allergan) injected intragastrically in the antrum every six months
  Other Names: Allergan

SUMMARY:
This is a pilot testing the feasibility of the 'REpurposing BOtulinum Toxin in Treatment of Obesity in Adolescents' trial (ReBOO-trial). The full-scale ReBOO will further investigate safety and efficacy of intragastric injections of botulinum toxin A into the antrum area of the stomach. These injections will be repeated every six months.

The study sample will be adolescents with obesity who have not responded to standard conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed) informed consent
2. Age and gender adjusted body mass index (ISO-BMI) ≥ 35 or ISO-BMI > 30 with comorbidities including hypertension, non-alcoholic fatty liver disease, hyperlipidemia or impaired glucose tolerance
3. Having partaken in a comprehensive multi-disciplinary lifestyle treatment for obesity of duration 12 months or more, without achieving a clinically significant weight loss (non-responder)

Exclusion Criteria:

1. Known hypersensitivity to excipients in the investigational medicine product (IMP)
2. Neuromuscular disorders
3. History of dysphagia
4. History of aspiration tendency or aspiration pneumonia
5. Known lung disease under continuous treatment
6. Congenital or acquired heart disease
7. Previous experience of side effects to Botulinum toxin type A
8. Present gastric diseases or dysfunction
9. Previous bariatric surgery
10. History of cancer
11. Serious binge eating disorder
12. Untreated hypothyroidism
13. Use of aminoglycoside antibiotics or spectinomycin in the week prior to injection, or any other medicinal product that interfere with neuromuscular transmission (neuromuscular blocking agents)
14. Medication known to affect appetite
15. Syndromic obesity
16. Mentally immature to a degree that there is doubt about the subject's ability to assent
17. Issues relating to language or culture that may complicate trial participation
18. Pregnancy or breastfeeding

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
BMI | 12 months
  Proportion of participants reaching a reduction in BMI z-score equal to or more than 1

SECONDARY OUTCOMES:
Injection interval | 12 months
  Patient reports will indicate the appropriate re-injection interval
Patient adherence to treatment | 12 months
  Qualitative data based on interviews with patients and next of kin.
Incidence of treatment-emergent adverse events | 2 years
  All adverse events (AE), serious adverse events (SAE) and suspected unexpected serious adverse reactions (SUSAR) will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Bård Eirik Kulseng, prof, Study Director — Norwegian University of Science and Technology, Fac MH, IKOM
Locations (1):
- St Olavs Hospital Trondheim University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No